CLINICAL TRIAL: NCT03559946
Title: A Randomized Controlled Trial Comparing the Efficacy of a Condensed (Twice Weekly) Protocol to the Standard (Once Per Week) Protocol of Percutaneous Tibial Nerve Stimulation (PTNS) in the Treatment of Overactive Bladder Syndrome (OAB)
Brief Title: Condensed Percutaneous Tibial Nerve Stimulation (PTNS) Protocol
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to COVID-19 pandemic
Sponsor: Stony Brook University (Other)
Collaborators: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Principal Investigator, Jason Kim, Clinical Assistant Professor of Urology, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1180838
Record Dates: First submitted 2018-06-08; First posted 2018-06-18 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Overactive Bladder Syndrome
Keywords: Overactive Bladder Syndrome; Percutaneous Tibial Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: We will be recruiting 66 patients, who will be randomized (1:1) to either the Standard Protocol (SP) group or the Condensed Protocol (CP) group.
Who Masked: Participant, Care Provider
Masking Description: Patients in both CP and SP groups will come to the clinic twice per week, and will not know their group assignment until the end of the study.
  All the interventions will be performed by the sub-investigator. The care providing physician will not know the group assignment of the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Protocol (SP) group (Sham Comparator): The patients in the SP group will receive one PTNS treatment and one sham treatment per week for 12 weeks
  Interventions: Device: percutaneous tibial nerve stimulation (PTNS); Device: Sham procedure
- Condensed Protocol (CP) group (Experimental): The patients in the CP group will receive 2 PTNS treatments per week for 12 weeks.
  Interventions: Device: percutaneous tibial nerve stimulation (PTNS)

INTERVENTIONS:
Device: percutaneous tibial nerve stimulation (PTNS) — The PTNS and the sham treatments will be given in 30 min sessions. The PTNS treatment consists of inserting a 34-gauge needle electrode approximately 5 cm cephalad to the medial malleolus and, as well as placing a PTNS surface electrode on the ipsilateral calcaneus. To keep the electrode placement consistent with the sham treatment, 2 inactive transcutaneous electrical nerve stimulation (TENS) surface electrodes are also added, 1 placed under the little toe and 1 on the top of the foot. The PTNS lead set is connected to the Urgent PC stimulator, and a current level of 0.5 to 10 mA at 20 Hz is delivered until the flexion of the big toe is observed or the patient reports a radiating sensation at the sole of the foot.
Device: Sham procedure — The sham treatment, involves simulating the sensation of the PTNS needle insertion at the same location using a Steritberger placebo needle. This is a blunt tip needle which simulates the sensation of a needle prick when touched to the skin, however, the blunt tip retracts into the handle when pressed into the skin. This creates the illusion of the needle entering the skin, without breaking the skin's surface. An inactive PTNS surface electrode is also placed on the ipsilateral calcaneus. The two TENS surface electrodes, placed in the same location as the PTNS treatment, are active and deliver stimulation mimicking the sensory effects of the PTNS. However, since no electrode needles were inserted near the tibial nerve, there will be no tibial nerve stimulation
  Arms: Standard Protocol (SP) group

SUMMARY:
The purpose of this study is to understand how the frequency of PTNS sessions impacts their efficacy in the treatment of over active bladder syndrome.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of the periodicity of the PTNS treatments on the efficacy of treating patients with OAB. We will compare the efficacy of a condensed (twice weekly) protocol to the standard (once per week) protocol of PTNS therapy.

Objective #1 (6-wk CP vs. 12-wk SP) is to show that 6 weeks of the condensed protocol (CP) will yield a higher efficacy compared to the standard 12-week protocol (SP). If this 6-week CP is proven effective, candidates for PTNS treatment could potentially experience symptom relief in half the time as the current standard of care, improving their quality of life quicker. Objective #2 (12-wk CP vs. 12-wk SP) is to show that 12 weeks of the CP will have a higher efficacy compared to the 12-week SP. If the superiority of this 12-week CP is proven, it could be beneficial in treating patients with refractory OAB.

ELIGIBILITY:
Inclusion Criteria:

* Women and men (18 years of age and older) with overactive bladder syndrome, who are interested in receiving PTNS treatment.

Exclusion Criteria:

* Patients with anatomical limitations preventing successful placement of the electrode, medical disorders precluding stimulation (bleeding disorders, cardiac pacemakers, peripheral vascular disease or ulcers, or lower leg cellulitis).
* Pregnant women or women who are planning to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Global Response Assessment (GRA) | At week 6 and week 12
  GRA asks the patents to rate how their urinary symptoms have changed since the start of the treatment on a 7-point scale (markedly worse, moderately worse, mildly worse, same, slightly improved, moderately improved, and markedly improved)

SECONDARY OUTCOMES:
Incontinence impact questionnaire-7 (IIQ-7) | At week 0, 6 and 12
  IIQ-7 contains 7 questions to assess how accidental urine loss has affected the patients' activities, relationships, and feelings.

OTHER OUTCOMES:
Urinary Distress Inventory (UDI) 6 short form | At week 0, 6 and 12
  UDI 6 contains 6 questions to assess the patients' urinary symptoms such as stress incontinence, urgency incontinence, frequency, pelvic pain and bladder emptying

CONTACTS AND LOCATIONS:
Overall Officials: Jason Kim, M.D., Principal Investigator — Stony Brook University Hospital, Department of Urology
Locations (1):
- Stony Brook Medicine Women's Pelvic Health And Continence Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peters KM, Carrico DJ, Perez-Marrero RA, Khan AU, Wooldridge LS, Davis GL, Macdiarmid SA. Randomized trial of percutaneous tibial nerve stimulation versus Sham efficacy in the treatment of overactive bladder syndrome: results from the SUmiT trial. J Urol. 2010 Apr;183(4):1438-43. doi: 10.1016/j.juro.2009.12.036. Epub 2010 Feb 20. PMID 20171677
- [Background] Finazzi-Agro E, Petta F, Sciobica F, Pasqualetti P, Musco S, Bove P. Percutaneous tibial nerve stimulation effects on detrusor overactivity incontinence are not due to a placebo effect: a randomized, double-blind, placebo controlled trial. J Urol. 2010 Nov;184(5):2001-6. doi: 10.1016/j.juro.2010.06.113. Epub 2010 Sep 20. PMID 20850833